CLINICAL TRIAL: NCT05342155
Title: Patient- Generated Health Data to Predict Childhood Cancer Survivorship Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HEALTHSHR; 1R01CA258193-01 (NIH)
Record Dates: First submitted 2022-03-08; First posted 2022-04-22 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Survivorship; Childhood Cancer
Keywords: Health Data
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Focus Group: For the focus group, the participant will be asked to review the potential platform the investigators are developing to better describe risks of health are developing to better describe risks of health issues in childhood cancer survivors. The focus group session will last approximately 2 hours.
- Campus and Home Assessments: For the campus and home assessments, the participant will be engaged in the research activities over 108 weeks (approximately 2 years).
  DatStat Connect app-Throughout participation in this research study, the participant will use a personal compatible device, such as smartphone or tablet, to report information about their health and respond to questionnaires using a website app called DatStat Connect.
  The wrist monitor (Actigraph) and heart monitor (CorSense) will also transmit information to DatStat Connect. The wrist monitor and heart monitor will connect to a compatible personal device via Bluetooth.
  The wrist monitor and heart CorSense device and St Jude Life study visit St Jude LIFE study visit: the participant will be asked to complete a St Jude LIFE research study assessment on the St Jude campus at three timepoints: initial visit (Week 0),approximately end of Year 1 (Week 60), and approximately end of Year 2 (Week 108).

SUMMARY:
Some childhood cancer survivors have health problems as the result of previous cancer treatment. This study is being done to determine if we can better predict the risk a childhood cancer survivor might have for developing future health issues.

The goal of this study is to enable regular monitoring of patient-generated health data (PGHD), including symptoms, physical activity, energy expenditure, sleep behavior and heart rate variability, and utilize these data in predicting survivor-specific risk of late effects to improve survivorship care and outcomes.

DETAILED DESCRIPTION:
This study is designed to collect symptoms/other PGHD as risk factors of subsequent adverse outcomes, including PROs (impaired QOL, unplanned healthcare use) assessed via smartphones, and clinical outcomes (physical performance deficits, onset of/worsening CHCs) assessed at SJCRH's After Completion of Therapy (ACT) Clinic. Each survivor will be assessed at 6 timepoints over 2-year period: T0 (baseline: week 0) for assessing baseline PROs and clinical outcomes at ACT Clinic; T1 (7 days in week 1), T2 (7 days in week 5) and T3 (7 days in week 9) for collecting symptoms/PGHD and PROs in non-clinical, daily-living settings; T4 (week 60) and T5 (week 108) for collecting PRO and clinical outcomes at ACT Clinic. Survivors will report symptoms/PGHD over a 3-month period for a purpose of collecting risk factors.

Primary Objective

Aim 1: Use a mHealth platform to collect and integrate symptoms, activity, and health behavioral data, and develop/validate risk prediction models for future QOL outcomes using these dynamic data.

Aim 1a: Investigate variability of patient-generated health data (PGHD), i.e., symptoms (via smartphone), and physical activity, energy expenditure, sleep behavior and heart rate variability (via wearable accelerometer/biometric sensor) within and between survivors with special attention to their temporal change patterns.

Aim 1b: Assess associations and temporal patterns of the mHealth-collected PGHD while considering clinical (cancer treatment exposure/doses, age at cancer diagnosis, childhood cancer types, etc.) and socio-demographic (age at study, sex, educational attainment, income, etc.) factors.

Aim 1c: Develop risk prediction models for future QOL outcomes using training data with cross-validation and validate model performance using independent test data.

Aim 1d: Establish personalized risk prediction scores for potential use within clinical settings.

Secondary Objectives

Aim 2: Develop/validate risk prediction models and establish personalized risk prediction scores for other outcomes (unplanned care utilization including emergency room visits and hospitalizations, physical performance deficits, onset of chronic health conditions) using the same approach as Aim 1.

Aim 3: Create a web-based tool to calculate and report personalized outcome specific risks and facilitate integration of risk scores into the survivor's patient portal and hospital's EHR for potential future use/evaluation in clinical management.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at the time of study
* Enrolled on SJLIFE
* ≥5 years from initial diagnosis of pediatric cancer/malignancy
* Currently not receiving cancer therapies
* Access to web-enabled smartphone

Exclusion Criteria:

* Known severe neurocognitive impairment (e.g., estimated intelligence score [FSIQ] <70), which requires proxies to complete daily symptom and PRO surveys;
* <3rd-grade reading level or not able to communicate in English;
* Currently pregnant or reports planning to become pregnant in the next two years;
* Lack of access to web-enabled smartphone, or not able to use/access internet from the device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants who meet eligibility criteria and consent to enrollment on the study
Sampling Method: Non-Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-20 (Estimated)

PRIMARY OUTCOMES:
Symptom log | Baseline, week 1, week 5, week 9, week 60 and week 108, timeline for each survivor includes 6 timepoints over 2-year period
  Log of patient reported symptoms
Euro QoL 5D | Baseline, week 1, week 5, week 9, week 60 and week 108, timeline for each survivor includes 6 timepoints over 2-year period
  Quality of Life Survey
NIH PROMIS 45 | Baseline, week 1, week 5, week 9, week 60 and week 108, timeline for each survivor includes 6 timepoints over 2-year period
  Patient report outcomes
QLACS | Baseline, week 1, week 5, week 9, week 60 and week 108, timeline for each survivor includes 6 timepoints over 2-year period
  Quality of Life in Adult Cancer Survivors Survey
MEPS-US Medical Expenditure Panel Survey | Baseline, week 1, week 5, week 9, week 60 and week 108, timeline for each survivor includes 6 timepoints over 2-year period
  Unplanned health care utilization (emergency room visits, hospitalization, unplanned primary care physician visit)
Chronic health conditions log | Baseline, week 60 and week 108
  Log of patient reported chronic health condition status
Physical performance-Cardiopulmonary fitness | Baseline , week 60 and week 108
  Cardiopulmonary fitness - six minute walk and cardiopulmonary exercise testing
Physical performance-Muscular strength and endurance | Baseline, week 60 and week 108
  Muscular strength and endurance - Isometric grip strength, isokinetic knee extension and ankle dorsiflexion (Biodex System 4)
Physical performance-Flexibility | Baseline, week 60 and week 108
  Flexibility - Sit and reach test (Flex-Tester), passive ankle range of motion
Physical performance-Mobility | Baseline, week 60 and week 108
  Mobility - Timed up and go test
Physical performance-Balance and sensory integrity | Baseline, week 60 and week 108
  Balance and sensory integrity - Computerized dynamic posturography (SMART Equi Test)

CONTACTS AND LOCATIONS:
Overall Officials: I-Chang Huang, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols